CLINICAL TRIAL: NCT02054104
Title: Adjuvant Tumor Lysate Vaccine and Iscomatrix With or Without Metronomic Oral Cyclophosphamide and Celecoxib in Patients With Malignancies Involving Lungs, Esophagus, Pleura, or Mediastinum
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Vaccine production halted in 2015, thus study is terminated.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, David Schrump, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 140053; 14-C-0053
Record Dates: First submitted 2014-02-01; First posted 2014-02-04 (Estimated); Results first posted 2022-01-26 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2021-12

CONDITIONS: Thoracic Sarcomas; Thorasic Cancers; Cancers of Non-thoracic Origin With Metastases to the Lungs or Pleura; Sarcoma; Melanoma
Keywords: Minimal Residual Disease; Cancer Vaccine; Immunotherapy; No Clinical Evidence of Active Disease
MeSH Terms: conditions — Sarcoma; Melanoma; Neoplasm, Residual | interventions — Cyclophosphamide; Celecoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1/Vaccine Plus Chemotherapy (Experimental): H1299 cell lysates with iscomatrix vaccine with metronomic chemotherapy
  Interventions: Biological: H1299 cell lysates; Drug: Cyclophosphamide; Drug: Celecoxib; Biological: Iscomatrix adjuvant
- 2/Vaccine Alone (Experimental): H1299 cell lysates with iscomatrix adjuvant vaccine
  Interventions: Biological: H1299 cell lysates; Biological: Iscomatrix adjuvant

INTERVENTIONS:
Biological: H1299 cell lysates — H1299 cell lysate with iscomatrix adjuvant vaccine via subcutaneous injections once every cycle (cycle=28 days) for 6 cycles total. Additional 2 injections for patients with immunologic response and no clinical evidence of active disease (NED).
Drug: Cyclophosphamide — 50 mg by mouth (PO) twice a day (BID) for 7 days prior to the first dose of vaccine and then on days 8 through 14, and 22 through 28 of each treatment cycle.
  Other Names: Cytoxan
  Arms: 1/Vaccine Plus Chemotherapy
Drug: Celecoxib — 400 mg by mouth (PO) twice a day (BID) for 7 days prior to the first dose of vaccine and then on days 1 through 28 of each treatment cycle.
  Other Names: Celebrex
  Arms: 1/Vaccine Plus Chemotherapy
Biological: Iscomatrix adjuvant — H1299 cell lysate with iscomatrix adjuvant vaccine via subcutaneous injections once every cycle (cycle=28 days) for 6 cycles total. Additional 2 injections for patients with immunologic response and no clinical evidence of active disease (NED).

SUMMARY:
Background:

During recent years, cancer-testis (CT) antigens (CTA), particularly those encoded by genes on the X chromosome (CT-X genes), have emerged as attractive targets for cancer immunotherapy. Whereas malignancies of diverse histologies express a variety of CTAs, immune responses to these proteins appear uncommon in cancer patients, possibly due to low-level, heterogeneous antigen expression, as well as immunosuppressive regulatory T cells present within tumor sites and systemic circulation of these individuals. Conceivably, vaccination of cancer patients with tumor cells expressing high levels of CTAs in combination with regimens that deplete or inhibit T regulatory cells will induce broad immunity to these antigens. In order to examine this issue, patients with primary lung and esophageal cancers, pleural mesotheliomas, thoracic sarcomas, thymic neoplasms and mediastinal germ cell tumors, as well as sarcomas, melanomas, germ cell tumors, or epithelial malignancies metastatic to lungs, pleura or mediastinum with no evidence of disease (NED) or minimal residual disease (MRD) following standard multidisciplinary therapy will be vaccinated with H1299 tumor cell lysates with Iscomatrix adjuvant. Vaccines will be administered with or without metronomic oral cyclophosphamide (50 mg by mouth (PO) twice a day (BID) x 7day (d) every (q) 14d), and celecoxib (400 mg PO BID). Serologic responses to a variety of recombinant CTAs as well as immunologic responses to autologous tumor or epigenetically modified autologous Epstein-Barr virus (EBV) transformed lymphocytes will be assessed before and after a six month vaccination period.

Primary Objectives:

1. To assess the frequency of immunologic responses to CTAs in patients with thoracic malignancies following vaccinations with H1299 cell lysate/Iscomatrix(TM) vaccines alone in comparison to patients with thoracic malignancies following vaccinations with H1299 cell lysate/Iscomatrix vaccines in combination with metronomic cyclophosphamide and celecoxib.

Secondary Objectives:

1. To examine if oral metronomic cyclophosphamide and celecoxib therapy diminishes the number and percentage of T regulatory cells and diminishes activity of these cells in patients with thoracic malignancies are at risk of recurrence.
2. To examine if H1299 cell lysate/Iscomatrix(TM) vaccination enhances immunologic response to autologous tumor or epigenetically modified autologous EBV-transformed lymphocytes (B cells).

Eligibility:

* Patients with histologically or cytologically proven small cell or non-small cell lung cancer (SCLC;NSCLC), esophageal cancer (EsC), malignant pleural mesothelioma (MPM), thymic or mediastinal germ cell tumors, thoracic sarcomas, or melanomas, sarcomas, or epithelial malignancies metastatic to lungs, pleura or mediastinum who have no clinical evidence of active disease (NED), or minimal residual disease (MRD) not readily accessible by non-invasive biopsy or resection/radiation following standard therapy completed within the past 26 weeks.
* Patients must be 18 years or older with an Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 2.
* Patients must have adequate bone marrow, kidney, liver, lung and cardiac function.
* Patients may not be on systemic immunosuppressive medications at time vaccinations commence.

Design:

* Following recovery from surgery, chemotherapy, or chemo/radiotherapy (XRT), patients with NED or MRD will be vaccinated via IM injection with H1299 cell lysates and Iscomatrix(TM) adjuvant monthly for 6 months.
* Vaccines will be administered with or without with metronomic oral cyclophosphamide and celecoxib.
* Systemic toxicities and immunologic response to therapy will be recorded. Pre and post vaccination serologic and cell mediated responses to a standard panel of CT antigens as well as autologous tumor cells (if available) and EBV-transformed lymphocytes will be assessed before and after vaccination.
* Numbers/percentages and function of T regulatory cells in peripheral blood will be assessed before, during, and after vaccinations.
* Patients will be followed in the clinic with routine staging scans until disease recurrence.
* The trial will randomize 28 evaluable patients per arm to either receive vaccine alone or vaccine plus chemotherapy in order to have 80% power to determine if the frequency of immune responses on the combination arm exceeds that of the vaccine alone arm, if the expected frequencies of immune responses on the two arms were 20% and 50%, using a one-sided 0.10 alpha level Fisher's exact test.
* Approximately 60 patients will be accrued to this trial.

DETAILED DESCRIPTION:
Background:

During recent years, cancer-testis (CT) antigens (CTA), particularly those encoded by genes on the X chromosome (CT-X genes), have emerged as attractive targets for cancer immunotherapy. Whereas malignancies of diverse histologies express a variety of CTAs, immune responses to these proteins appear uncommon in cancer patients, possibly due to low-level, heterogeneous antigen expression, as well as immunosuppressive regulatory T cells present within tumor sites and systemic circulation of these individuals. Conceivably, vaccination of cancer patients with tumor cells expressing high levels of CTAs in combination with regimens that deplete or inhibit T regulatory cells will induce broad immunity to these antigens. In order to examine this issue, patients with primary lung and esophageal cancers, pleural mesotheliomas, thoracic sarcomas, thymic neoplasms and mediastinal germ cell tumors, as well as sarcomas, melanomas, germ cell tumors, or epithelial malignancies metastatic to lungs, pleura or mediastinum with no evidence of disease (NED) or minimal residual disease (MRD) following standard multidisciplinary therapy will be vaccinated with H1299 tumor cell lysates with Iscomatrix (Trademark) adjuvant. Vaccines will be administered with or without metronomic oral cyclophosphamide (50 mg by mouth (PO) twice a day (BID) x 7day (d) every (q) 14d), and celecoxib (400 mg PO BID). Serologic responses to a variety of recombinant CTAs as well as immunologic responses to autologous tumor or epigenetically modified autologous Epstein-Barr Virus (EBV) transformed lymphocytes will be assessed before and after receiving 6 vaccines.

Primary Objectives:

-To assess the frequency of immunologic responses to CTAs in patients with thoracic malignancies following vaccinations with H1299 cell lysate/Iscomatrix (Trademark) vaccines alone in comparison to patients with thoracic malignancies following vaccinations with H1299 cell lysate/Iscomatrix (Trademark) vaccines in combination with metronomic cyclophosphamide and celecoxib.

Eligibility:

-Patients with histologically or cytologically proven small cell or non-small cell lung cancer (SCLC;NSCLC), esophageal cancer (EsC), malignant pleural mesothelioma (MPM), thymic or mediastinal germ cell tumors, thoracic sarcomas, or melanomas, sarcomas, or

epithelial malignancies metastatic to lungs, pleura or mediastinum who have no clinical evidence of active disease (NED), or minimal residual disease (MRD) not readily accessible by non-invasive biopsy or resection/radiation following standard therapy completed within the past 56 weeks.

* Patients must be 18 years or older with an Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 2.
* Patients must have adequate bone marrow, kidney, liver, lung and cardiac function.
* Patients may not be on systemic immunosuppressive medications at time vaccinations commence.

Design:

* Following recovery from surgery, chemotherapy, or chemo/XRT, patients with NED or MRD will be vaccinated via deep subcutaneous (SQ) injection with H1299 cell lysates and Iscomatrix (Trademark) adjuvant monthly until 6 vaccinations have been given.
* Vaccines will be administered with or without with metronomic oral cyclophosphamide and celecoxib.
* Systemic toxicities and immunologic response to therapy will be recorded. Pre and post vaccination serologic and cell mediated responses to a standard panel of CT antigens as well as autologous tumor cells (if available) and EBV-transformed lymphocytes will be assessed before and after vaccination.
* Numbers/percentages and function of T regulatory cells in peripheral blood will be assessed before, during, and after vaccinations.
* Patients will be followed in the clinic with routine staging scans until disease recurrence.
* The trial will randomize 28 evaluable patients per arm to either receive vaccine alone or vaccine plus chemotherapy in order to have 80% power to determine if the frequency of immune responses on the combination arm exceeds that of the vaccine alone arm, if the expected frequencies of immune responses on the two arms were 20% and 50%, using a one-sided 0.10 alpha level Fisher's exact test.
* Approximately 60 patients will be accrued to this trial.

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Patients with histologically or cytologically proven lung or esophageal cancers, thymic or mediastinal germ cell tumors, malignant pleural mesotheliomas, or primary thoracic sarcomas, as well as patients with sarcomas, melanomas, germ cell tumors, or epithelial malignancies metastatic to the lungs, mediastinum, or pleura that have no clinical evidence of active disease (NED) or minimal residual disease (MRD) not readily accessible by non-invasive biopsy or resection/radiation following standard therapy.
2. Diagnosis must be confirmed by the National Cancer Institute (NCI) Laboratory of Pathology.
3. Patients must be enrolled within 56 weeks following completion of therapy.
4. Patients must have completed standard therapy for their malignancy and recovered from all toxicities to less than or equal to Grade 2 within 3 weeks prior to enrollment.
5. Patients with intracranial metastases, which have been treated by surgery or radiation therapy, may be eligible for study provided there is no evidence of active disease and no requirement for anticonvulsant therapy or steroids following treatment.
6. Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 2
7. Patients must be 18 years of age or older due to the unknown effects of immunologic responses to this vaccine during childhood and adolescent development.
8. Patients must have evidence of adequate bone marrow reserve, hepatic and renal function as evidenced by the following laboratory parameters:

   * Absolute neutrophil count greater than 1500/mm^3
   * Platelet count greater than 100,000/mm^3
   * Hemoglobin greater than 8g/dl (patients may receive transfusions to meet this parameter)
   * Prothrombin (PT) within 2 seconds of the upper limit of normal (ULN)
   * Total bilirubin <1.5 x upper limits of normal
   * Serum creatinine less than or equal to 1.6 mg/ml or the creatinine clearance must be greater than 70 ml/min/1.73m^2.
9. Seronegative for human immunodeficiency virus (HIV) antibody. Note: The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who are HIV seropositive may have decreased immune competence and thus may be less responsive to the experimental treatment.
10. Seronegative for active hepatitis B, and seronegative for hepatitis C antibody. If hepatitis C antibody test is positive, then patient must be tested for the presence of antigen by reverse transcription polymerase chain reaction (RT-PCR) and be hepatitis C virus (HCV) ribonucleic acid (RNA) negative.
11. The effects of the study treatment on the developing human fetus are unknown; thus, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) within 28 days prior to study entry, for the duration of study participation and up to 120 days after the last dose of the drug. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
12. Patients must be willing to sign an informed consent.
13. Ability and willingness to co-enroll on the screening and tissue collection protocol 06C0014, 'Prospective Evaluation of Genetic and Epigenetic Alterations in Patients with Thoracic Malignancies'.

EXCLUSION CRITERIA:

1. Patients who are initially rendered no clinical evidence of active disease (NED) or have minimal residual disease (MRD) following standard therapy but exhibit disease progression prior to initiation of vaccination will be excluded from the study.
2. Patients requiring chronic systemic treatment with steroids will be excluded.
3. Patients receiving warfarin anticoagulation, who cannot be transitioned to other agents such as enoxaparin or dabigatran, and for whom anticoagulants cannot be held for up to 24 hours will be excluded.
4. Patients with uncontrolled hypertension (>160/95), unstable coronary disease evidenced by uncontrolled arrhythmias, unstable angina, decompensated congested heart failure (CHF) (>New York Heart Association (NYHA) Class II), or myocardial infarction within 6 months of study will be excluded.
5. Patients with other cardiac diseases may be excluded at the discretion of the PI following consultation with Cardiology consultants.
6. Patients with any of the following pulmonary function abnormalities will be excluded: forced expiratory volume (FEV), < 30% predicted; carbon monoxide (DLCO) < 30% predicted (post-bronchodilator); oxygen saturation less than 92% on room air.
7. Female patients who are pregnant or breastfeeding. Because there is unknown, potentially harmful effects of immune response to CT-X antigens and stem cell proteins that may be expressed in placenta, fetus, and neonates.
8. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations 3 months prior to enrollment that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2014-09-03 (Actual); Primary Completion 2015-06-03 (Actual); Study Completion 2015-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David S Schrump, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schrump DS. Targeting epigenetic mediators of gene expression in thoracic malignancies. Biochim Biophys Acta. 2012 Jul;1819(7):836-45. doi: 10.1016/j.bbagrm.2012.03.009. Epub 2012 Apr 9. PMID 22507242
- [Background] Cheng YH, Wong EW, Cheng CY. Cancer/testis (CT) antigens, carcinogenesis and spermatogenesis. Spermatogenesis. 2011 Jul-Sep;1(3):209-220. doi: 10.4161/spmg.1.3.17990. Epub 2011 Jul 1. PMID 22319669
- [Background] Fratta E, Coral S, Covre A, Parisi G, Colizzi F, Danielli R, Nicolay HJ, Sigalotti L, Maio M. The biology of cancer testis antigens: putative function, regulation and therapeutic potential. Mol Oncol. 2011 Apr;5(2):164-82. doi: 10.1016/j.molonc.2011.02.001. Epub 2011 Feb 18. PMID 21376678
- [Result] Zhang M, Hong JA, Kunst TF, Bond CD, Kenney CM, Warga CL, Yeray J, Lee MJ, Yuno A, Lee S, Miettinen M, Ripley RT, Hoang CD, Gnjatic S, Trepel JB, Schrump DS. Randomized phase II trial of a first-in-human cancer cell lysate vaccine in patients with thoracic malignancies. Transl Lung Cancer Res. 2021 Jul;10(7):3079-3092. doi: 10.21037/tlcr-21-1. PMID 34430349
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2014-C-0053.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1/Vaccine Plus Chemotherapy: H1299 cell lysates with iscomatrix vaccine with metronomic chemotherapy
  H1299 cell lysates: H1299 cell lysate with iscomatrix adjuvant vaccine via subcutaneous injections once every cycle (cycle=28 days) for 6 cycles total. Additional 2 injections for patients with immunologic response and no clinical evidence of active disease (NED).
  Cyclophosphamide: 50 mg by mouth (PO) twice a day (BID) for 7 days prior to the first dose of vaccine and then on days 8 through 14, and 22 through 28 of each treatment cycle.
  Celecoxib: 400 mg by mouth (PO) twice a day (BID) for 7 days prior to the first dose of vaccine and then on days 1 through 28 of each treatment cycle.
  Iscomatrix adjuvant: H1299 cell lysate with iscomatrix adjuvant vaccine via subcutaneous injections once every cycle (cycle=28 days) for 6 cycles total. Additional 2 injections for patients with immunologic response and no clinical evidence of active disease (NED).
- Cohort 2/Vaccine Alone: H1299 cell lysates with iscomatrix adjuvant vaccine
  H1299 cell lysates: H1299 cell lysate with iscomatrix adjuvant vaccine via subcutaneous injections once every cycle (cycle=28 days) for 6 cycles total. Additional 2 injections for patients with immunologic response and no clinical evidence of active disease (NED).
  Iscomatrix adjuvant: H1299 cell lysate with iscomatrix adjuvant vaccine via subcutaneous injections once every cycle (cycle=28 days) for 6 cycles total. Additional 2 injections for patients with immunologic response and no clinical evidence of active disease (NED).
Period: Overall Study
Arm/Group | Cohort 1/Vaccine Plus Chemotherapy | Cohort 2/Vaccine Alone
Started | 10 | 11
Completed | 2 | 2
Not Completed | 8 | 9
Not completed — Did not want to continue due to college classes | 1 | 0
Not completed — Biopsy positive for malignancy, appears to be new primary | 1 | 0
Not completed — No evidence of immunologic response | 2 | 2
Not completed — Disease Progression On Study | 4 | 5
Not completed — Diagnosis of lymphoma | 0 | 1
Not completed — Inconclusive response | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1/Vaccine Plus Chemotherapy | Cohort 2/Vaccine Alone | Total
Number analyzed (Participants) | 10 | 11 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 8 | 17
  >=65 years | 1 | 3 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.48 (16.96) | 48.59 (17.82) | 47.59 (17.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 5 | 7 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 8 | 11 | 19
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 8 | 10 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 10 | 11 | 21

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With an Immunologic Responses
Description: Immunologic responses are defined as an appearance of new serologic reactivity, or increase in existing antibody response to cancer-testis on the X chromosome (CT-X) antigen. Antigens such as New York esophageal squamous cell carcinoma-1 (NY-ESO1) and melanoma antigen gene (MAGE) family members assessed by enzyme-linked immunosorbent assay (ELISA) one month after the 6th vaccine.
Time Frame: one month after the 6th vaccine
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1/Vaccine Plus Chemotherapy | Cohort 2/Vaccine Alone
Number analyzed (Participants) | 10 | 11
Participants | 4 | 4

2. Secondary Outcome: Fold Change From Baseline of Intensity of Programmed Cell Death Protein 1(PD-1) Expression on Tregs
Description: The Mann=Whitney U test was used to compare the fold change of intensity of PD-1 expression on Tregs between the two groups. A decrease in the fold change is consistent with a better outcome. The difference, or the relative difference, in the values at the two time points were obtained and tested to determine if the difference is equal to zero. If a paired t-test is able to be used, with at least 20 evaluable participants, there is 81% power to detect a change equal to ¾ of a standard deviation of the change at the two-sided 0.025 significance level. This was done in order to allow for a conservative adjustment due to determining the significance of the change in the percent of Tregs on two arms.
Time Frame: one month after first 6 vaccinations
Measure: Mean (Full Range); unit: fold change
Arm/Group | Cohort 1/Vaccine Plus Chemotherapy | Cohort 2/Vaccine Alone
Number analyzed (Participants) | 7 | 7
fold change | 0.84 [0.67 to 1.07] | 0.91 [0.79 to 1.03]

3. Secondary Outcome: Fold Change From Baseline of Percent Tregs
Description: The Mann-Whitney U test was used to compare the fold change of percent Tregs between the two groups. A decrease in the fold change is consistent with a better outcome. The difference, or the relative difference, in the values at the two time points were obtained and tested to determine if the difference is equal to zero. If a paired t-test is able to be used, with at least 20 evaluable participants, there is 81% power to detect a change equal to ¾ of a standard deviation of the change at the two-sided 0.025 significance level. This was done in order to allow for a conservative adjustment due to determining the significance of the change in the percent of Tregs on two arms.
Time Frame: one month after first 6 vaccinations
Measure: Mean (Full Range); unit: fold change
Arm/Group | Cohort 1/Vaccine Plus Chemotherapy | Cohort 2/Vaccine Alone
Number analyzed (Participants) | 7 | 7
fold change | 0.87 [0.65 to 1.12] | 0.73 [0.23 to 1.13]
Statistical Analysis 1: Comparison: Cohort 1/Vaccine Plus Chemotherapy vs Cohort 2/Vaccine Alone; Test type: Other; p = 0.36, Mann-Whitney U test

4. Other Pre Specified Outcome: Percentage of T Regulatory Cells at the Two Timepoints: Baseline and End of Treatment
Description: The immunologic response to autologous tumor or epigenetically-modified autologous Epstein-Barr Virus (EBV)-transformed lymphocytes will be determined by the difference, or relative difference, in values (by percentage) of T-regulatory cells at the two timepoints. The percentage of T-regulatory cells will determine if oral cyclophosphamide and celecoxib therapy decreases the percentage of T cells on each Arm/Group.
Time Frame: Baseline, and end of treatment
Population: This exploratory endpoint was not assessed because the trial was suspended after only 1/3rd of the total anticipated patient accrual.
Arm/Group | Cohort 1/Vaccine Plus Chemotherapy | Cohort 2/Vaccine Alone
Number analyzed (Participants) | 0 | 0

5. Other Pre Specified Outcome: Number of Participants With Serious and Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0)
Description: Here is the number of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to final collection of AE data, approximately 9 months and 12 days for cohort 1 and 8 months and 22 days for cohort 2.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1/Vaccine Plus Chemotherapy | Cohort 2/Vaccine Alone
Number analyzed (Participants) | 10 | 11
Participants | 8 | 6

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to final collection of AE data, approximately 9 months and 12 days for cohort 1 and 8 months and 22 days for cohort 2.
Arm/Group | Cohort 1/Vaccine Plus Chemotherapy | Cohort 2/Vaccine Alone
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/11
Other Adverse Events (participants affected / at risk) | 8/10 | 6/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1/Vaccine Plus Chemotherapy (N=10) | Cohort 2/Vaccine Alone (N=11)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
CPK increased (Investigations) | 2 (2) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 1 (2)
Flu like symptoms (General disorders) | 1 (1) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 2 (4)
Lymphocyte count decreased (Investigations) | 7 (16) | 3 (5)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 3 (6) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
White blood cell decreased (Investigations) | 5 (8) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-03): https://cdn.clinicaltrials.gov/large-docs/04/NCT02054104/Prot_SAP_000.pdf
  • Informed Consent Form (2021-04-14): https://cdn.clinicaltrials.gov/large-docs/04/NCT02054104/ICF_001.pdf